CLINICAL TRIAL: NCT05698030
Title: Efficacy of Oral Immunotherapy to Pistachio in Children on the Oral Tolerance to Pistachio and Cashew Nuts
Brief Title: Efficacy and Saffety of Oral Immunotherapy to Pistachio
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Amandine DIVARET-CHAUVEAU, MCU-PH, Central Hospital, Nancy, France
Other Study IDs: 2022PI182
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Allergy; Food Allergy
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Food allergy — Oral immunotherapy to pistachio

SUMMARY:
The objectives of this study are (i) to evaluate the efficacy of oral immunotherapy to pistachio by evaluating the daily oral tolerance of 2g pistachio, by evaluating the long-term tolerance of 15g pistachio (sustained unresponsiveness) and by decreasing pistachio-specific IgE, (ii) evaluating the efficacy of pistachio immunotherapy on cashew tolerance, (iii) and to evaluate the safety of pistachio immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years of age with a proven allergy to pistachio and followed in the pediatric allergology unit of the Nancy University Hospital.
* Patients who have received oral immunotherapy to pistachio for at least 18 months at 31/12/2022

Exclusion Criteria:

* Patients who have received oral immunotherapy to pistachio for less than 18 months.
* Patients lost to follow-up for more than 2 years or last consultation dating from 2020 or earlier

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients meeting the inclusion criteria (between 10 and 50)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Absence of moderate to severe allergic reactions | during the 6 months of maintenance
  with daily intake of 2g of pistachio

SECONDARY OUTCOMES:
Frequency and severity of allergic reactions | during the dose escalation phase and during the maintenance phase (first 6 months, 1st year, 2nd year, 3rd year)
Decrease in specific IgE and increase of IGg4 to pistachio | during the dose escalation phase and during the maintenance phase (first 6 months, 1st year, 2nd year, 3rd year)
Tolerance of 1, 2, 4, 8g in isolated doses and 15 g in total cumulative dose of pistachio | 3 months after stopping daily consumption of 2g pistachio
  during an oral pistachio challenge test
Tolerance of 1, 2, 4, 8g in isolated doses and 15 g in total cumulative dose of cashew nut | 3 months after stopping daily consumption of 2g pistachio
  during an oral cashew nut challenge test
Reactogenic or tolerogenic threshold of cashew nuts | during the dose escalation phase and during the maintenance phase (first 6 months, 1st year, 2nd year, 3rd year)

CONTACTS AND LOCATIONS:
Overall Officials: Amandine DIVARET-CHAUVEAU, Principal Investigator — Centre hospitalo-universitaire de Nancy
Locations (1):
- Centre Hospitalo-Universitaire de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No